CLINICAL TRIAL: NCT05123222
Title: Phase I Evaluation of Two Zika Viruses for Use in Controlled Human Infection Models (CHIM)
Brief Title: Evaluation of Two Zika Viruses for Use in Controlled Human Infection Models (CHIM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIR 316
Record Dates: First submitted 2021-10-26; First posted 2021-11-17 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Zika Virus
Keywords: Zika virus
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Intervention Model Description: This study will include 4 cohorts of 14 ZIKV and DENV-naïve non-pregnant female and male subjects, 18 - 40 years of age (total: 56 subjects). Within each cohort, 10 subjects will receive ZIKV and 4 subjects will receive a placebo on Study Day 0. Cohorts 1 and 2 (Dose = 10^2 PFU) will be enrolled first and will enroll only women. Cohorts 3 and 4 (Dose = 10^2 PFU) will enroll men. Two strains of ZIKV will be evaluated in both men and women- San Jose Rio Puerto (Cohorts 1 and 3) and Nicaragua (Cohorts 2 and 4).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - SJRP (Experimental): ZIKV-SJRP/2016-184 injected at dose of 10^2 PFU.
  Interventions: Biological: ZIKV-SJRP/2016-184 Strain
- Cohort 1 - Placebo (Placebo Comparator): Volume matched placebo injection (saline)
  Interventions: Biological: Placebo
- Cohort 2 - Nicaragua (Experimental): ZIKV-Nicaragua/2016 injected at dose of 10^2 PFU.
  Interventions: Biological: Experimental: ZIKV-Nicaragua/2016 Strain
- Cohort 2 - Placebo (Placebo Comparator): Volume matched placebo injection (saline)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ZIKV-SJRP/2016-184 Strain — Zika Virus Strain (San Jose Rio Puerto)
  Arms: Cohort 1 - SJRP
Biological: Experimental: ZIKV-Nicaragua/2016 Strain — Zika Virus Strain (Nicaragua)
  Arms: Cohort 2 - Nicaragua
Biological: Placebo — Saline
  Arms: Cohort 1 - Placebo; Cohort 2 - Placebo

SUMMARY:
This study will include 4 cohorts of 14 ZIKV and DENV-naïve female and male subjects, 18 - 40 years of age (total: up to 56 subjects). Within each cohort, 10 subjects will receive ZIKV and 4 subjects will receive a placebo on Study Day 0. Cohorts 1 and 2 (Dose = 10^2 PFU) will be enrolled first and will enroll only women. Cohorts 3 and 4 (Dose = 10^2 PFU) will enroll men.

DETAILED DESCRIPTION:
This study is a placebo-controlled, double-blind study in normal healthy adult male and non-pregnant female subjects 18 - 40 years of age, inclusive, recruited from the metropolitan Baltimore/Washington, DC and Burlington, VT areas. The purpose of this study is to evaluate the clinical and virologic response to escalating doses of 2 different ZIKV strains administered subcutaneously in healthy, ZIKV and DENV-naïve, male and non-pregnant, female adult volunteers to identify the most suitable ZIKV strain and dose for use in a ZIKV CHIM. The ZIKV CHIM will then be used to evaluate the protective efficacy of candidate ZIKV vaccines prior to evaluation of these candidates in Phase 2 clinical trials. Both ZIKV strains will be studied at doses of 10^2 PFU. Placebo recipients are included in the study as a control to better assess ZIKV-associated versus non-ZIKV-associated AEs.

ELIGIBILITY:
Inclusion Criteria:

* Adult ZIKV and DENV-naïve male and non-pregnant females 18 - 40 years of age, inclusive.
* Good general health as determined by physical examination, laboratory screening, and review of medical history.
* Available for the duration of the study, approximately 26 weeks post-inoculation.
* Must be able to complete the informed consent process and comprehension assessment independently and without assistance.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Willingness to reside in the inpatient unit for 9 days (or longer for safety if necessary) following receipt of ZIKV or placebo.
* Male subjects: Willingness to use barrier contraception during cervico-vaginal, anal, and oral intercourse through study day 90 (in accordance with CDC guidance).
* Female subjects: Willingness to use barrier contraception during cervico-vaginal, anal, and oral intercourse through study day 56 (in accordance with CDC guidance).
* Female subjects of childbearing potential must be willing to use effective contraception while at risk of Zika infection. CDC guidelines for the use of effective contraception of 8 weeks post-infection will be followed; time of infection is defined as inoculation with challenge virus. Reliable methods of contraception include: hormonal birth control* (implantable, hormonal patch, hormonal vaginal ring, oral contraception, Depo-Provera injection, etc.), surgical sterilization (hysterectomy, tubal ligation, or tubal coil at least 3 months prior to inoculation), and intrauterine device. All female subjects will be considered having child-bearing potential except for those with post-menopausal status documented as at least 1 year since last menstrual period and females who have sex with females (exclusively) and have no intention of conceiving a child during the study. Females who are not considered to be of childbearing potential will not be required to use contraception other than barrier contraception for the purpose of reducing potential transmission.

  * Volunteers on hormonal birth control must not be on medications or other agents that decrease the effectiveness of hormonal birth control.

Exclusion Criteria:

* Currently pregnant, as determined by positive beta-human choriogonadotropin (Beta-hCG) test, breast-feeding or planning to become pregnant during the 6-month duration of the study.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the requirements of the study protocol.
* Evidence of recent opiate use based on urine toxicology screen
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), ALT, and serum creatinine, as defined in this protocol.
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by subject history.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (emergency room visit or hospitalization within the last 6 months).
* HIV infection, by screening and confirmatory assays.
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays.
* Hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening.
* History of Guillain-Barré syndrome (GBS).
* History of seizure disease or peripheral neuropathy
* History of any neuroinflammatory disorder i.e. Bell's Palsy, transverse myelitis
* Any known immunodeficiency syndrome, including that caused by malignancy.
* Use of anticoagulant medications (use of antiplatelet medication such as aspirin or non-steroidal anti-inflammatory medication is permitted and will not exclude a subject from enrollment).
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following inoculation. Immunosuppressive dose of corticosteroids is defined as ≥10 mg prednisone equivalent per day for ≥14 days.
* Receipt of a live vaccine within 21 days or a killed vaccine within the 14 days prior to inoculation or anticipated receipt of any vaccine during the 21 days following inoculation.
* Asplenia.
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following inoculation.
* History or serologic evidence of previous ZIKV infection or DENV infection.
* Previous receipt of a ZIKV or DENV vaccine (licensed or investigational).
* Anticipated receipt of any investigational agent in the 28 days before or after inoculation.
* Subject has definite plans to travel to a ZIKV-endemic or dengue-endemic area during the study.
* Previous hypersensitivity to any study product component.
* Anaphylactic reaction to mosquito bites.
* Refusal to allow storage of specimens for future research.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ZIKV-SJRP/2016-184 Strain: Dose of 10ˆ2 PFU
  ZIKV-SJRP/2016-184 Strain: Zika Virus Strain (San Jose Rio Puerto)
- ZIKV-SJRP/2016-184 Strain Placebo; ZIKV-Nicaragua/2016 Strain Placebo: Volume matched placebo injection (saline)
- ZIKV-Nicaragua/2016 Strain: Dose of 10ˆ2 PFU
  Experimental: ZIKV-Nicaragua/2016 Strain: Zika Virus Strain (Nicaragua)
Period: Overall Study
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016-184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Started | 20 | 8 | 20 | 8
Completed | 18 | 8 | 19 | 8
Not Completed | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ZIKV-SJRP/2016-184 Strain: ZIKV-SJRP/2016-184 at dose 10^2 PFU.
- ZIKV-SJRP/2016-184 Strain Placebo; ZIKV-Nicaragua/2016 Strain Placebo: Volume-matched placebo injection (saline).
- ZIKV-Nicaragua/2016 Strain: ZIKV-Nicaragua/2016 at dose 10^2 PFU.
- Total: Total of all reporting groups
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016-184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo | Total
Number analyzed (Participants) | 20 | 8 | 20 | 8 | 56
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0 | 0 | 0
  18-50 | 20 | 8 | 20 | 8 | 56
  >=51 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 10 | 4 | 28
  Male | 10 | 4 | 10 | 4 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 2 | 10 | 1 | 21
  White | 9 | 4 | 6 | 5 | 24
  More than one race | 2 | 1 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 8 | 20 | 8 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Solicited Adverse Events
Description: measured by count of solicited adverse events recorded following ZIKV administration
Time Frame: Through 90 days post-inoculation
Measure: Number; unit: events
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016-184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 20 | 8 | 20 | 8
events
  Injection Site Erythema | 1 | 0 | 0 | 0
  Injection Site Tenderness | 2 | 1 | 3 | 1
  Injection Site Pain | 0 | 0 | 0 | 0
  Injection Site Pruritus | 0 | 0 | 0 | 0
  Injection Site Induration | 0 | 0 | 0 | 0
  Fever | 0 | 0 | 0 | 0
  Headache | 48 | 8 | 42 | 17
  Zika-like Rash | 21 | 2 | 29 | 2
  Neutropenia | 2 | 0 | 2 | 0
  Nonpurulent Conjunctivitis | 6 | 0 | 6 | 1
  Myalgia | 13 | 0 | 16 | 2
  Arthralgia | 13 | 2 | 12 | 0
  Retro-orbital Pain | 6 | 0 | 14 | 3
  Fatigue | 17 | 4 | 21 | 4
  Muscle Weakness | 1 | 0 | 0 | 0
  Hyporeflexia | 0 | 0 | 0 | 0
  Thrombocytopenia | 0 | 0 | 0 | 0
  Leukopenia | 2 | 0 | 7 | 0
  Pruritus | 4 | 0 | 1 | 1
  Photophobia | 5 | 1 | 7 | 0

2. Primary Outcome: Severity of Adverse Events
Description: count of solicited AEs by severity grade 1 - mild, event that is easily tolerated, may require 1 dose of medication.
  grade 2 - moderate, event that interferes with daily activity or requires more than 1 dose of medication.
  grade 3 - severe, event that prevents daily activity and requires medical intervention.
  grade 4 - life-threatening, an adverse event that is deemed by the study clinician, the medical monitor, or an outside clinician caring for the subject to be a life-threatening event.
  grade 5 - death, any adverse event that results in the death of the subject.
Time Frame: Through 90 days post-inoculation
Measure: Number; unit: events
Groups:
- ZIKV-SJRP/2016-184 Strain: ZIKV-SJRP/2016 injected at dose of 10^2 PFU.
- ZIKV-SJRP/2016_184 Strain Placebo; ZIKV-Nicaragua/2016 Strain Placebo: Volume matched placebo injection (saline)
- ZIKV-Nicaragua/2016 Strain: ZIKV-Nicaragua/2016 injected at dose of 10^2 PFU.
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016_184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 20 | 8 | 20 | 8
events
  Grade 1 | 181 | 47 | 212 | 45
  Grade 2 | 34 | 8 | 38 | 7
  Grade 3 | 0 | 1 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Infected by ZIKV
Description: Infection defined as recovery of ZIKV by RT-PCR from blood and/or by seroconversion to ZIKV (50% plaque reduction neutralization titer [PRNT50]≥ 1:10)
Time Frame: Through 90 days post-inoculation
Measure: Count of Participants; unit: Participants
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016-184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 20 | 8 | 20 | 8
Participants | 20 | 0 | 20 | 0

4. Primary Outcome: Number of Participants With Zika Virus Recovered From Serum, Whole Blood, CVS, Semen, Urine, and Saliva
Description: Count of participants with infectious virus recovered from serum, whole blood, cervicovaginal secretions (CVS), semen, urine, and saliva as measured by RT-PCR
Time Frame: Through 90 days post-inoculation
Population: Only participants infected by ZIKV. CVS was collected from female participants and semen was collected from male participants.
Measure: Count of Participants; unit: Participants
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016_184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 20 | 0 | 20 | 0
Participants
  Serum | 20 |  | 20 |
  Whole blood | 20 |  | 20 |
  Cervicovaginal secretions: number analyzed (Participants) | 10 | 0 | 10 | 0
  Cervicovaginal secretions | 6 |  | 7 |
  Semen: number analyzed (Participants) | 10 | 0 | 10 | 0
  Semen | 4 |  | 7 |
  Urine | 10 |  | 7 |
  Saliva | 8 |  | 7 |

5. Primary Outcome: Magnitude of ZIKV Recovered From Serum, Whole Blood, CVS, Semen, Urine, and Saliva
Description: Mean peak titer of ZIKV recovered in serum, whole blood, cervicovaginal secretions (cvs), semen, urine, and saliva of participants by RT-PCR. Data are reported in Log10 Genome Equivalents (GE) per milliliter.
Time Frame: Through 90 days post-inoculation
Population: Only participants from whom infectious virus was recovered. The number analyzed per specimen type is the number of participants from whom infectious virus was recovered. CVS was collected from female participants and semen was collected from male participants.
Measure: Mean (Standard Error); unit: log10GE/mL
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016_184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 20 | 0 | 20 | 0
log10GE/mL
  Serum | 5.27 (0.10) |  | 6.26 (0.10) |
  Whole blood | 4.46 (0.11) |  | 5.54 (0.11) |
  CVS: number analyzed (Participants) | 6 | 0 | 7 | 0
  CVS | 3.28 (0.50) |  | 3.17 (0.46) |
  Semen: number analyzed (Participants) | 4 | 0 | 7 | 0
  Semen | 5.94 (1.0) |  | 5.22 (0.76) |
  Urine: number analyzed (Participants) | 10 | 0 | 7 | 0
  Urine | 3.54 (0.38) |  | 3.32 (0.46) |
  Saliva: number analyzed (Participants) | 8 | 0 | 7 | 0
  Saliva | 2.72 (0.20) |  | 2.84 (0.22) |

6. Primary Outcome: Duration of ZIKV in Serum, Whole Blood, CVS, Semen, Urine, and Saliva
Description: Mean number of days that ZIKV was recovered in serum, whole blood, cervicovaginal secretions (cvs), semen, urine, and saliva from participants with detectable zika as measured by RT-PCR
Time Frame: Through 90 days post-inoculation
Population: as for outcome 5
Measure: Mean (Standard Error); unit: days
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016_184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 20 | 0 | 20 | 0
days
  Serum | 7.3 (0.47) |  | 8.1 (0.48) |
  Whole Blood | 7.0 (0.52) |  | 6.2 (0.52) |
  Cervicovaginal secretions: number analyzed (Participants) | 6 | 0 | 7 | 0
  Cervicovaginal secretions | 3.3 (0.93) |  | 4.4 (0.86) |
  Semen: number analyzed (Participants) | 4 | 0 | 7 | 0
  Semen | 7.3 (3.39) |  | 13.0 (2.57) |
  Urine: number analyzed (Participants) | 10 | 0 | 7 | 0
  Urine | 3.1 (0.96) |  | 3.6 (1.15) |
  Saliva: number analyzed (Participants) | 8 | 0 | 7 | 0
  Saliva | 2.6 (1.02) |  | 2.7 (1.10) |

7. Secondary Outcome: Frequency of AEs by Severity
Description: Number of AEs by grade grade 1 - mild, event that is easily tolerated, may require 1 dose of medication.
  grade 2 - moderate, event that interferes with daily activity or requires more than 1 dose of medication.
  grade 3 - severe, event that prevents daily activity and requires medical intervention.
  grade 4 - life-threatening, an adverse event that is deemed by the study clinician, the medical monitor, or an outside clinician caring for the subject to be a life-threatening event.
  grade 5 - death, any adverse event that results in the death of the subject.
Time Frame: Through 28 days post-inoculation
Measure: Number; unit: events
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016_184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 20 | 8 | 20 | 8
events
  Grade 1 | 179 | 46 | 211 | 44
  Grade 2 | 32 | 7 | 34 | 5
  Grade 3 | 0 | 1 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Zika Virus Recovered From Serum, Whole Blood, CVS, Semen, Urine, and Saliva
Description: determined by number of participants with infectious virus in serum, whole blood, cervicovaginal secretions (cvs), semen, urine, and saliva as measured by virus culture
Time Frame: Through 90 days post-inoculation
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016_184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 20 | 0 | 20 | 0
Participants
  Serum | 20 |  | 20 |
  Whole Blood | 14 |  | 18 |
  CVS: number analyzed (Participants) | 10 | 0 | 10 | 0
  CVS | 1 |  | 1 |
  Semen: number analyzed (Participants) | 10 | 0 | 10 | 0
  Semen | 5 |  | 4 |
  Urine | 3 |  | 2 |
  Saliva | 7 |  | 14 |

9. Secondary Outcome: Peak Virus Titer Recovered From Serum, Whole Blood, CVS, Semen, Urine, and Saliva
Description: mean peak titer of ZIKV in participants with ZIKV recovered from serum, whole blood, cervicovaginal secretions (cvs), semen, urine, and saliva by virus culture. Data are reported in Log10 Genome Equivalents (GE) per milliliter.
Time Frame: Through 90 days post-inoculation
Population: Only participants from whom infectious virus was recovered. The number analyzed per specimen type is the number of participants from whom infectious virus was recovered. CVS was collected for female participants and semen was collected for male participants.
Measure: Mean (Standard Error); unit: log10GE/mL
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016_184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 20 | 0 | 20 | 0
log10GE/mL
  Serum | 2.12 (0.17) |  | 3.65 (0.14) |
  Whole Blood: number analyzed (Participants) | 14 | 0 | 18 | 0
  Whole Blood | 2.20 (0.11) |  | 3.57 (0.10) |
  CVS: number analyzed (Participants) | 1 | 0 | 1 | 0
  CVS | 2.30 |  | 2.70 |
  Semen: number analyzed (Participants) | 5 | 0 | 4 | 0
  Semen | 3.67 (0.81) |  | 3.87 (0.91) |
  Urine: number analyzed (Participants) | 3 | 0 | 2 | 0
  Urine | 1.19 (0.24) |  | 1.0 (0.29) |
  Saliva: number analyzed (Participants) | 7 | 0 | 14 | 0
  Saliva | 0.96 (0.23) |  | 1.01 (0.17) |

10. Secondary Outcome: Duration of ZIKV in Serum, Whole Blood, CVS, Semen, Urine, and Saliva
Description: mean number of days that ZIKV was recovered in serum, whole blood, cervicovaginal secretions (cvs), semen, urine, and saliva from participants with detectable zika as measured by virus culture
Time Frame: Through 90 days post-inoculation
Population: as for outcome 5
Measure: Mean (Standard Error); unit: days
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016_184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 20 | 0 | 20 | 0
days
  Serum | 4.8 (0.24) |  | 5.0 (0.24) |
  Whole blood: number analyzed (Participants) | 14 | 0 | 18 | 0
  Whole blood | 2.8 (0.38) |  | 3.9 (0.34) |
  CVS: number analyzed (Participants) | 1 | 0 | 1 | 0
  CVS | 1.0 |  | 3.0 |
  semen: number analyzed (Participants) | 5 | 0 | 4 | 0
  semen | 3.6 (1.4) |  | 6.0 (1.57) |
  urine: number analyzed (Participants) | 3 | 0 | 2 | 0
  urine | 1.7 (0.54) |  | 1.0 (0.67) |
  saliva: number analyzed (Participants) | 7 | 0 | 14 | 0
  saliva | 2.1 (0.77) |  | 3.0 (0.54) |

11. Secondary Outcome: Peak Neutralizing Antibody Response to ZIKV
Description: evaluate the kinetics of the serum neutralizing antibody response following primary ZIKV infection.
Time Frame: Through 90 days post-inoculation
Population: participants with at least 1 measurement during the 90-day time period are included in the analysis
Measure: Mean (Standard Error); unit: log10GE/mL
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016_184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
Number analyzed (Participants) | 18 | 0 | 20 | 0
log10GE/mL | 6129 (0) |  | 4265 (0) |

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | ZIKV-SJRP/2016-184 Strain | ZIKV-SJRP/2016-184 Strain Placebo | ZIKV-Nicaragua/2016 Strain | ZIKV-Nicaragua/2016 Strain Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/8 | 0/20 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/8 | 0/20 | 1/8
Other Adverse Events (participants affected / at risk) | 20/20 | 8/8 | 20/20 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZIKV-SJRP/2016-184 Strain (N=20) | ZIKV-SJRP/2016-184 Strain Placebo (N=8) | ZIKV-Nicaragua/2016 Strain (N=20) | ZIKV-Nicaragua/2016 Strain Placebo (N=8)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZIKV-SJRP/2016-184 Strain (N=20) | ZIKV-SJRP/2016-184 Strain Placebo (N=8) | ZIKV-Nicaragua/2016 Strain (N=20) | ZIKV-Nicaragua/2016 Strain Placebo (N=8)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 5 (9) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (18) | 3 (4) | 6 (10) | 0 (0)
Insomnia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (2) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (5) | 0 (0)
Dysmenorrhea (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Venipuncture site bruise (General disorders) | 1 (1) | 3 (3) | 8 (11) | 2 (2)
AST increased (Hepatobiliary disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 6 (11) | 0 (0) | 7 (9) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (4)
Back pain (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 4 (5) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Application site pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 4 (4) | 2 (2)
Injection site tenderness (General disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 16 (48) | 5 (8) | 16 (42) | 5 (17)
Zika-like rash (Skin and subcutaneous tissue disorders) | 17 (21) | 2 (2) | 20 (29) | 1 (2)
Leukopenia (Immune system disorders) | 2 (2) | 0 (0) | 6 (7) | 0 (0)
Non-purulent conjunctivitis (Eye disorders) | 6 (6) | 0 (0) | 6 (6) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
ALT increased (Hepatobiliary disorders) | 4 (4) | 3 (8) | 3 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (13) | 0 (0) | 13 (16) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 1 (2) | 9 (12) | 0 (0)
Photophobia (Eye disorders) | 3 (4) | 1 (1) | 4 (7) | 0 (0)
Retro-orbital pain (Eye disorders) | 5 (6) | 0 (0) | 8 (14) | 2 (3)
Fatigue (General disorders) | 10 (17) | 4 (4) | 14 (22) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiatal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Immune system disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Muscle ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Light headedness (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Common cold (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flu (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dog bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Belching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergic rhinitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Night sweats (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT05123222/Prot_SAP_000.pdf